CLINICAL TRIAL: NCT06087016
Title: Urinary Markers by SpectrosCopy: Diagnostic Aid in oncologY - Application to Urological Cancer
Brief Title: Urinary Markers by SpectrosCopy: Diagnostic Aid in oncologY - Application to Urological Cancers
Acronym: MUSCADE
Status: Recruiting | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO23014
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Urinary Bladder Tumour
Keywords: URINARY BLADDER NEOPLASMS; DIAGNOSIS; URINE; ANALYSIS; Spectroscopy; Fourier Transform Infrared; Raman; Spectrum Analysis; Multivariate Analysis
MeSH Terms: conditions — Urinary Bladder Neoplasms; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bladder cancer group: Bladder cancer group represents patients attending or hospitalized in Urology department, Reims University Hospital and in whom, tumor is visualized during cystoscopy and confirmed by the histological examination of entire resected lesion after Trans Urethral Resection of Bladder Tumor (TURBT).
  Interventions: Other: Urine vibrational analysis
- Control group: Control group includes patients consulting for cystoscopy examination in Urology department, Reims University Hospital without any tumor visualization during cystoscopy examination.
  Interventions: Other: Urine vibrational analysis

INTERVENTIONS:
Other: Urine vibrational analysis — Urine vibrational analysis

SUMMARY:
This study aims to evaluate the performance of vibrational spectroscopy (Infrared and Raman spectroscopy techniques) in bladder cancer diagnosis using urine samples.

DETAILED DESCRIPTION:
Urologic cancers affect the organs and structures of the male and female urinary tract and the male reproductive system. Bladder cancer (BCa) is the second urological cancer in incidence after prostate cancer and represents the 10th most common cancer in the world. This cancer has high recurrence and progression rates. Cystoscopy and urine cytology are the current gold-standard examination for bladder cancer. Nevertheless, the first is invasive and the latter has low sensitivity especially for low-grade bladder cancer. Therefore, it is critical to implement accurate, non- invasive and sensitive examination tool to diagnose patients with bladder cancer at an early stage.

On the one hand, urine is collected non-invasively and considered as a proximal biofluid from bladder. On the other hand, vibrational spectroscopy including Infrared and Raman spectroscopy is widely used for the analysis of biological samples and provides a molecular fingerprint of the sample with minimum or no sample preparation. Applied on urine, this technique may offer interesting alternative for bladder cancer diagnosis and monitoring. Hence, this research project aims to evaluate the analytical capabilities of urinary vibrational spectroscopy with the objective of developing a diagnostic test for urothelial bladder cancer.

The study is planned for 36 months. Patients that approve their participation in the study will respond to a questionnaire allowing us to have clinical information. From these patients, urine samples will be collected in Urology department of Reims University Hospital. Urine samples will be directly analyzed by Fourier Transform Infrared Spectroscopy and/or Surface-enhanced Raman spectroscopy then stored at -80°C for further analysis.

ELIGIBILITY:
inclusion criteria:

* Must be over 18 years of age
* Able to give consent and understand the purpose the study
* Agree to participate in the study and having signed the non-objection document
* Admitted to a urology consultation for cystoscopy

exclusion criteria: Patients with any of the following criteria will not be included in the study

* Refused to participate in the study or unable to give consent
* without a native bladder
* with a bladder fistula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending for cystoscopy examination or hospitalized in Urology department, Reims University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2025-03-06 (Estimated); Study Completion 2026-03-06 (Estimated)

PRIMARY OUTCOMES:
Fourier Transform Infrared Spectroscopy | A 36 months
  Analyze urine samples by infrared spectroscopy after drying step and without any further sample preparation. The obtained spectra will be preprocessed and analyzed by multivariate algorithms to discriminate bladder cancer patients from control group.

SECONDARY OUTCOMES:
Surface-enhanced Raman spectroscopy | A 36 months
  Analyze urine samples by Surface-enhanced Raman spectroscopy after mixing urine samples with silver nanoparticles. The obtained spectra will be preprocessed and analyzed by multivariate algorithms to discriminate bladder cancer patients from control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France